CLINICAL TRIAL: NCT04062539
Title: Total Cerebral Protection With Embolic Protection Devices in Thoracic Aortic Stenting
Brief Title: Total Cerebral Protection With Embolic Protection Devices Thoracic Aortic Stenting
Status: Suspended | Type: Observational
Why Stopped: Waiting for funding
Sponsor: Imperial College London (Other)
Collaborators: St Mary's Hospital, London (Other)
Responsible Party: Sponsor
Other Study IDs: INTERCEPT:CEPD
Record Dates: First submitted 2019-04-12; First posted 2019-08-20 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Stroke; Silent Cerebral Infarct
Keywords: stroke; cerebral embolic protection device
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All captured material from the filters will be analysed and this can include atherosclerotic particles and thrombus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Sentinel and Spider — Dual filter and single filter

SUMMARY:
Stroke and silent cerebral infarction are a real risk with thoracic enodvascular aortic repair (TEVAR). The investigator propose to prospectively observational study with enrolment of all patients undergoing TEVAR for thoracic and thoracoabdominal conditions including aneurysmal degeneration, Type B dissection and acute aortic syndromes over a 24 month period, equating to a minimum of 20-30 patients per year. Patients undergoing juxtra-renal and infra-renal aortic stenting will form a control group.

DETAILED DESCRIPTION:
TEVAR involves the insertion of a stent into the thoracic aorta to re-line it and prevent life-threatening haemorrhage from rupture, and ultimately death. The stent is inserted through a small cut in the femoral artery in the groin that is able to track to the desired location in the thoracic aorta over wires. The thoracic aorta and the branches it provides to supply the brain are diseased with atherosclerotic plaques and thrombus. The manipulation of wires and stents over these diseased locations can lead to small fragments breaking off and travelling to the brain to block the blood supply to areas of the brain (cerebral embolisation).

Cerebral embolic protection devices (CEPDs) consist of filters that can be placed into the branches of the thoracic aorta that supply the brain(supra-aortic branches) before TEVAR and can capture and remove solid debris, preventing it from reaching the brain.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring TEVAR as decided upon by a multidisciplinary meeting

Exclusion Criteria:

* Contraindication to MRI scanning
* Unable to give consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Secondary care; elective patients from an outpatient clinical bases and emergency patients presenting through Accident and Emergency
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of brain injury assessed by Magnetic resonance imaging (MRI) test | Pre-operative and post-operative up to 6 months
  Magnetic resonance imaging (MRI) of the brain is a safe and painless test that uses a magnetic field and radio waves to produce detailed images of the brain.

SECONDARY OUTCOMES:
Incidence of embolic event | Intra-operative
  Transcranial doppler monitoring of embolic events
Changes in neurocognition function | Pre-operative and post-operative up until 6 months
  Neurocognitive tests to assess the changes in neurocognition function

CONTACTS AND LOCATIONS:
Overall Officials: Richard Gibbs, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perera AH, Rudarakanchana N, Monzon L, Bicknell CD, Modarai B, Kirmi O, Athanasiou T, Hamady M, Gibbs RG. Cerebral embolization, silent cerebral infarction and neurocognitive decline after thoracic endovascular aortic repair. Br J Surg. 2018 Mar;105(4):366-378. doi: 10.1002/bjs.10718. Epub 2018 Feb 12. PMID 29431856
- [Background] Grover G, Perera AH, Hamady M, Rudarakanchana N, Barras CD, Singh A, Davies AH, Gibbs R. Cerebral embolic protection in thoracic endovascular aortic repair. J Vasc Surg. 2018 Dec;68(6):1656-1666. doi: 10.1016/j.jvs.2017.11.098. Epub 2018 May 24. PMID 29804744